CLINICAL TRIAL: NCT05791825
Title: Cultivating Healthy Intentional Mindful Educators (CHIME): The Use of Mindfulness and Compassion to Promote Early Head Start/Head Start Education Staffs Well-Being
Brief Title: Evaluation of the CHIME Intervention for Improving Early Head Start/Head Start Educator Well-being
Acronym: CHIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska Lincoln (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22130
Record Dates: First submitted 2023-02-13; First posted 2023-03-30 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Health, Subjective; Work Related Stress; Compassion; Social Skills
Keywords: Mindfulness; Social-emotional learning; Self-compassion; Early care and education; Teacher well-being; Head Start
MeSH Terms: conditions — Occupational Stress; Social Skills

STUDY DESIGN:
Intervention Model Description: The study employs a cluster-randomized design with two study arms, one of which will receive the intervention and the other of which will act as the control group. The study will employ repeated measures at pre- (baseline/time 1 assessment), post-intervention (time 2), and 3-month (time 3) follow-up points. The counterfactual will be a waitlisted control comparison condition and randomization to the intervention/control group will occur at the classroom level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receives CHIME (Experimental): Half of the educators participating in the trial will be assigned to this condition. CHIME is an 8-week, mindfulness and self-compassion based intervention that teaches educators strategies to enhance socioemotional learning in the classroom. The primary endpoints are: educator mindfulness and self-compassion, educator emotional regulation, educator heart rate variability, educator wellbeing and socio-emotional learning, and educator responsiveness, support, and sensitivity in the classroom. The secondary endpoints are: child self-regulation and social skills and family-school relationships.
  Interventions: Behavioral: Cultivating Healthy Intentional Mindful Educators
- Wait-listed comparison (No Intervention): Half of the HS/EHS educators will be assigned to a waitlisted control group. Specifically, these educators will be scheduled to receive the intervention after a 6-month waiting period. During the interim period, they will complete the same assessments as Arm 1, but will continue to receive 'business as usual' support and professional development through typical Head Start/EHS programming.

INTERVENTIONS:
Behavioral: Cultivating Healthy Intentional Mindful Educators — The 8-week, manualized, CHIME intervention consists of a 2-hour overview and seven weekly sessions, each lasting 90 minutes. Each CHIME session focuses on a specific mindfulness technique, such as mindful breathing, mindful listening and bringing attention to current states and surroundings to support optimal responsiveness, emotion regulation, and compassion. Social emotional learning is promoted by focusing on five broad competencies: self-awareness, social awareness, responsible decision-making, self-management, and relationship skills and these competencies are practiced and developed through small group discussions, storytelling, journal reflections, modeling, and guided awareness (e.g., meditations), and implementation activities (e.g., gratitude necklace).
  Arms: Receives CHIME

SUMMARY:
This study will test how well a mindfulness-based intervention called CHIME improves the emotional well-being of educators in Early Head Start and Head Start (EHS/HS) settings. The study also will examine if there are any benefits to young children's social emotional health as a result of the CHIME program. Researchers will compare educators who participate in CHIME to educators who are asked to participate at a later time to see if there are benefits to their emotional health and teaching practices.

DETAILED DESCRIPTION:
To address the critical need of supporting Early Head Start/Head Start (EHS/HS) education staff well-being, investigators are collaborating with EHS/HS programs to co-refine and adapt a new mindfulness-based intervention (MBI), Cultivating Healthy Intentional Mindful Educators (CHIME-HS), to make the intervention effective and internally sustainable for EHS/HS programs. Small studies with CHIME in general early care and education settings provide a proof of concept of its effectiveness, with educators reporting enhanced well-being and reduced workplace burnout. However, CHIME has not been adapted for or rigorously tested in EHS/HS settings. Building on promising evidence for the efficacy of CHIME, investigators partnered with EHS/HS programs to gather feedback from EHS and HS staff and families about how to refine CHIME to best address their needs, and determine CHIME's feasibility, acceptability, and fidelity within the EHS/HS context. In this way, investigators will maximize CHIME's acceptability, feasibility, and sustainability specifically for the unique needs of the HS/EHS start community. Investigators draw upon tenets of community-engaged research to co-refine and adapt the program to address EHS/HS education staff's well-being more effectively, and with sustainability in mind. After investigators refine CHIME in phase 1, investigators will work with EHS/HS partners to coordinate a rigorous, multi-method approach to evaluate the efficacy of CHIME with 120 EHS/HS education staff and 730 children/families (Phase 2). Investigators will also interview 10 directors and assistant EHS/HS directors to identify barriers and facilitators to implementation and to put in place effective mechanisms to support the sustainability of CHIME-HS (Phase 3). Through the iterative development and refinement of the facilitator training, investigators will determine if trained EHS/HS staff can effectively implement CHIME with fidelity for promoting EHS/HS education staff emotional well-being and workplace engagement, decreasing their physiological and emotional reactivity, promoting positive teaching practices, strengthening family partnerships, and promoting young children's social skills and self-regulation. Additionally, investigators will engage with other Early Head Start/Head Start University Partnership (HSUP) grantees during the yearly grantee workshop to share lessons learned, identify opportunities for collaborative analyses, and create shared dissemination products. A variety of dissemination efforts will be utilized to make findings from the study accessible to multiple audiences invested in EHS and HS populations. Dissemination products will include the CHIME-HS intervention, its promise for improving education staff well-being, outcomes, and lessons learned about implementation, including usability, feasibility, and cost. Investigators will work cooperatively with the consortium to disseminate policy findings recognizing that collective presentation and publication of findings can concentrate the impact.

ELIGIBILITY:
Inclusion Criteria:

There are 3 types of participants included in this study: Early Head Start/Head Start education staff who work at one of the partner sites; parents of children attending EHS or HS; children attending EHS or HS and enrolled in the classroom of a participating EHS/HS educator.

Inclusion criteria for each of these groups are as follows:

Early Head Start and Head Start Educators:

* Provision of signed and dated informed consent form in Docusign
* Currently employed as a lead or assistant educator for >20 hours per week in a participating Head Start or Early Head Start center
* Stated intention to participate in the CHIME intervention
* All genders; age 19 and older
* Able to complete activities in English

Parents

* Provision of electronically (in Docusign) /manually signed informed consent form
* All genders
* Age 19 and older
* is Parent or legal guardian of child enrolled in the classroom of a EHS/HS educator participating in the study
* Able to complete activities

Children

* Provision of electronically signed informed consent form by parent/legal guardian
* All genders; aged < 6 years
* Enrolled in the classroom of a EHS/HS educator participating in the study
* If > 3 years, ability to complete study activities in English or with translation support

Exclusion Criteria:

Exclusion criteria for each of the study groups are as follows:

Early Head Start and Head Start Educators:

* Does not currently work at a participating HS/EHS center
* younger than 19 years of age

Parents

* Not a parent/legal guardian of a child in an EHS/HS classroom
* younger than 19 years of age Children NA, although children less than 3 years will not complete the self-regulation tasks These exclusion criteria are essential to the design of the study. The population of interest is EHS/HS education staff (e.g., teachers) working within centers that have agreed to participate in the evaluation of CHIME. The legal age of majority in Nebraska is age 19 years.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Teacher Emotion Regulation Difficulties from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  Difficulties in Emotion Regulation Scale
Change in Teacher Adaptive Emotion Regulation from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  Emotion Regulation Questionnaire - Reappraisal scale
Change in Teacher Self-Compassion from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  Self-Compassion Scale
Change in Teacher Workplace Stress from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  NIOSH Worker Wellbeing Questionnaire
Change in Teacher Mental Well-Being from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  Warkwick-Edinburgh Mental Wellbeing Scale measures perceptions of overall mental well-being
Change in Educator heart rate variability from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  Actihearts worn in the classroom
Change in Teacher Depressive Symptoms from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  Center for Epidemiological Depression - Short From measuring depressive symptoms
Change Teaching Practices from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  Educator scores on the CLASS Observation Emotional Support Scale measuring the teachers emotional support for all the children in the classroom
Change in Teaching Practices from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  Caregiver Interaction Scale that measures the interactions between the participating educator and a target child in the classroom.

SECONDARY OUTCOMES:
Change in Child Social Skills from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  Child Social Skills Improvement System Socio-Emotional Learning Brief that measures social-emotional competencies
Change in Child Self-Regulation Skills from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  child self-regulation task scores from a puppet task administered with a trained researcher
Change in Perceived Family and Teacher Relationships from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  a measure of tahe quality of the relationship between the main primary caregiver and the teacher/educator) (Family and Provider Relationship Quality; Kim, 2012)
Change in Child Social Skills from baseline to post assessments | Baseline, a post-assessment 8 weeks after the intervention or waitlist period, and a follow-up assessment after 3 months.
  Devereux Early Childhood Assessment which is a behavior rating scale that is completed by parents and/or caregivers or teachers which provides an assessment of within-child protective factors central to social and emotional health and resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Hatton-Bowers, PhD, Principal Investigator — University of Nebraska Lincoln
Locations (1):
- University of Nebraska-Lincoln, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] Alvares GA, Quintana DS, Hickie IB, Guastella AJ. Autonomic nervous system dysfunction in psychiatric disorders and the impact of psychotropic medications: a systematic review and meta-analysis. J Psychiatry Neurosci. 2016 Mar;41(2):89-104. doi: 10.1503/jpn.140217. PMID 26447819
- [Background] Beauchaine TP. Respiratory Sinus Arrhythmia: A Transdiagnostic Biomarker of Emotion Dysregulation and Psychopathology. Curr Opin Psychol. 2015 Jun 1;3:43-47. doi: 10.1016/j.copsyc.2015.01.017. PMID 25866835
- [Background] Brody GH, Dorsey S, Forehand R, Armistead L. Unique and protective contributions of parenting and classroom processes to the adjustment of African American children living in single-parent families. Child Dev. 2002 Jan-Feb;73(1):274-86. doi: 10.1111/1467-8624.00405. PMID 14717257
- [Background] Chari R, Chang CC, Sauter SL, Petrun Sayers EL, Cerully JL, Schulte P, Schill AL, Uscher-Pines L. Expanding the Paradigm of Occupational Safety and Health: A New Framework for Worker Well-Being. J Occup Environ Med. 2018 Jul;60(7):589-593. doi: 10.1097/JOM.0000000000001330. PMID 29608542
- [Background] Dewhirst, C., & Goldman, J. (2018). Launching motivation for mindfulness: Introducing mindfulness to early childhood preservice teachers. Early Child Development and Care, 1-14, Advance online publication.. https://doi.org/10.1080/03004430.2018.1531853.
- [Background] Hamre BK, Pianta RC. Can instructional and emotional support in the first-grade classroom make a difference for children at risk of school failure? Child Dev. 2005 Sep-Oct;76(5):949-67. doi: 10.1111/j.1467-8624.2005.00889.x. PMID 16149994
- [Background] Hatton-Bowers H, Clark C, Parra G, Calvi J, Bird MY, Avari P, Foged J, Smith J. Promising Findings that the Cultivating Healthy Intentional Mindful Educators' Program (CHIME) Strengthens Early Childhood Teachers' Emotional Resources: An Iterative Study. Early Child Educ J. 2022 Aug 8:1-14. doi: 10.1007/s10643-022-01386-3. Online ahead of print. PMID 35967911
- [Background] Hays RD, Schalet BD, Spritzer KL, Cella D. Two-item PROMIS(R) global physical and mental health scales. J Patient Rep Outcomes. 2017;1(1):2. doi: 10.1186/s41687-017-0003-8. Epub 2017 Sep 12. PMID 29757325
- [Background] Holmes C, Levy M, Smith A, Pinne S, Neese P. A Model for Creating a Supportive Trauma-Informed Culture for Children in Preschool Settings. J Child Fam Stud. 2015;24(6):1650-1659. doi: 10.1007/s10826-014-9968-6. PMID 25972726
- [Background] Lomas T, Medina JC, Ivtzan I, Rupprecht S, Eiroa-Orosa FJ. A systematic review of the impact of mindfulness on the well-being of healthcare professionals. J Clin Psychol. 2018 Mar;74(3):319-355. doi: 10.1002/jclp.22515. Epub 2017 Jul 28. PMID 28752554
- [Background] Mackrain, M., LeBuffe, P. A., & Powell, G. (2007). The Devereux Early Childhood Assessment for Infants and Toddlers (DECA-I/T) assessment, technical manual, and user's guide. Lewisville, NC: Kaplan.
- [Background] Neff, K. D. (2003). The development and validation of a scale to measure self-compassion. Self and Identity, 2, 223-250. https://doi.org/10.1080/15298860309027
- [Background] Paniccia M, Paniccia D, Thomas S, Taha T, Reed N. Clinical and non-clinical depression and anxiety in young people: A scoping review on heart rate variability. Auton Neurosci. 2017 Dec;208:1-14. doi: 10.1016/j.autneu.2017.08.008. Epub 2017 Aug 26. PMID 28870754
- [Background] Perry, D., Allen, M. D., Brennan, E. M., & Bradley, J. R. (2010). The evidence base for mental health consultation in early childhood settings: A research synthesis addressing children's behavioral outcomes. Early Education & Development, 21, 795-824.
- [Background] Pianta, R. C. (2001). The Student-Teacher Relationship Scale. Lutz, FL: PAR.
- [Background] Pianta, R. C., Clifford, R., Burchinal, M., Bryant, D., Clifford, R., Early, D., & Barbarin, O. A. (2005). Features of pre-kindergarten programs, classrooms, and teachers: Do they predict observed classroom quality and child-teacher interactions. Applied Developmental Science, 9, 144-159. https://doi.org/10.1207/s1532480xads0903
- [Background] Porges, S. W., & Lewis, G. F. (2010). The polyvagal hypothesis: Common mechanisms mediating autonomic regulation, vocalizations and listening. In S. M. Burdzynski (Ed.), Handbook of Behavioral Neuroscience (Vol. 19, pp. 255-264). https://doi.org/10.1016/B978-0-12-374593-4.00025-5
- [Background] Santor, D. a., & Coyne, J. C. (1997). Shortening the CES-D to improve its ability to detect cases of depression. Psychological Assessment, 9(3), 233-243. https://doi.org/10.1037/1040-3590.9.3.233
- [Background] Schmitt, T. A. (2011). Current methodological considerations in exploratory and confirmatory factor analysis. Journal of Psychoeducational Assessment, 29, 4, 304-321.
- [Background] Shearer, A., Hunt, M., Chowdhury, M., & Nicol, L. (2015). Effects of a brief mindfulness meditation intervention on student stress and heart rate variability. International Journal of Stress Management, 23, 232-254. https://doi.org/10.1037/a0039814
- [Background] Yin H, Huang S, Wang W. Work Environment Characteristics and Teacher Well-Being: The Mediation of Emotion Regulation Strategies. Int J Environ Res Public Health. 2016 Sep 13;13(9):907. doi: 10.3390/ijerph13090907. PMID 27649216
- [Background] Zinsser KM, Christensen CG, Torres L. She's supporting them; who's supporting her? Preschool center-level social-emotional supports and teacher well-being. J Sch Psychol. 2016 Dec;59:55-66. doi: 10.1016/j.jsp.2016.09.001. Epub 2016 Oct 4. PMID 27923441
- [Background] Williams JM, Mathews A, MacLeod C. The emotional Stroop task and psychopathology. Psychol Bull. 1996 Jul;120(1):3-24. doi: 10.1037/0033-2909.120.1.3. PMID 8711015
- [Background] Ziv Y. Social information processing patterns, social skills, and school readiness in preschool children. J Exp Child Psychol. 2013 Feb;114(2):306-20. doi: 10.1016/j.jecp.2012.08.009. Epub 2012 Oct 6. PMID 23046690
- [Background] Park G, Van Bavel JJ, Vasey MW, Thayer JF. Cardiac vagal tone predicts attentional engagement to and disengagement from fearful faces. Emotion. 2013 Aug;13(4):645-56. doi: 10.1037/a0032971. PMID 23914769